CLINICAL TRIAL: NCT02965456
Title: A Phase 3, Multi-Center, Randomized, Double-Blind, Vehicle-Controlled, 2-Arm, Parallel Group Comparison Study Comparing the Efficacy and Safety of IDP-121 and IDP-121 Vehicle Lotion in the Treatment of Acne Vulgaris
Brief Title: Efficacy and Safety of IDP-121 and IDP-121 Vehicle Lotion in the Treatment of Acne Vulgaris
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: V01-121A-302
Record Dates: First submitted 2016-10-11; First posted 2016-11-16 (Estimated); Results first posted 2019-12-18 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Acne
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IDP-121 Lotion (Experimental): IDP-121 lotion (tretinoin 0.05 percent [%]) will be applied topically to the face of participants with moderate to severe acne, once daily for 12 weeks.
  Interventions: Drug: IDP 121 Lotion
- IDP-121 Vehicle Lotion (Placebo Comparator): IDP-121 lotion vehicle will be applied topically to the face of participants with moderate to severe acne, once daily for 12 weeks.
  Interventions: Drug: IDP-121 Vehicle Lotion

INTERVENTIONS:
Drug: IDP 121 Lotion — IDP-121 lotion will be applied as per the instructions provided by the investigational center staff.
  Arms: IDP-121 Lotion
Drug: IDP-121 Vehicle Lotion — IDP-121 vehicle lotion will be applied as per the instructions provided by the investigational center staff.
  Arms: IDP-121 Vehicle Lotion

SUMMARY:
The objective of this study was to evaluate the efficacy, safety, and tolerability of a once daily topical application of IDP-121 Lotion compared with its vehicle (IDP-121 Vehicle Lotion) in participants with moderate to severe acne vulgaris (acne) (that is, acne having an Evaluator's Global Severity Score [EGSS] of 3 [moderate] or 4 [severe]).

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female at least 9 years of age and older.
* Written and verbal informed consent must be obtained. Participants less than age of consent must sign an assent for the study and a parent or a legal guardian must sign the informed consent (if participant reaches age of consent during the study they should be re-consented at the next study visit).
* Participants must be willing to comply with study instructions and return to the study center for required visits. Participants under the age of consent must be accompanied by the parent or legal guardian at the time of assent/consent signing.
* If a cleanser, moisturizer or sunscreen is needed during the study, participants must be willing to use only allowed cleansers, moisturizers, sunscreens, or moisturizer/sunscreen combination products. If the participant wears makeup they must agree to use non-comedogenic makeup.

Key Exclusion Criteria:

* Use of an investigational drug or device within 30 days of enrollment or participation in a research study concurrent with this study.
* Any dermatological conditions on the face that could interfere with clinical evaluations such as acne conglobata, acne fulminans, secondary acne, perioral dermatitis, clinically significant rosacea, gramnegative folliculitis.
* Any underlying disease(s) or some other dermatological condition of the face that requires the use of interfering topical or systemic therapy or makes evaluations and lesion count inconclusive.
* Participants with a facial beard or mustache that could interfere with the study assessments.
* History of hypersensitivity or allergic reactions to any of the study preparations as described in the Investigator's Brochure, including known sensitivities to any dosage form of tretinoin.
* Participants who are unable to communicate or cooperate with the Investigator due to language problems, poor mental development, or impaired cerebral function.
* Participants with any underlying disease that the Investigator deems uncontrolled, and poses a concern for the participant's safety while participating in the study.

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 820 (Actual)
Dates: Start 2015-11-04 (Actual); Primary Completion 2017-02-23 (Actual); Study Completion 2017-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim Theisen, Study Chair — TKL Research, Inc.
Locations (34):
- United States (34):
  - Valeant Site 21, Glendale, Arizona
  - Valeant Site 34, Rogers, Arkansas
  - Valeant Site 25, Anaheim, California
  - Valeant Site 18, Beverly Hills, California
  - Valeant Site 09, Fremont, California
  - Valeant Site 17, Murrieta, California
  - Valeant Site 26, Oxnard, California
  - Valeant Site 22, Sacramento, California
  - Valeant Site 02, San Diego, California
  - Valeant Site 04, San Diego, California
  - Valeant Site 19, Santa Monica, California
  - Valeant Site 15, Miami, Florida
  - Valeant Site 11, Miami, Florida
  - Valeant Site 27, Pinellas Park, Florida
  - Valeant Site 31, Sanford, Florida
  - Valeant Site 05, Tampa, Florida
  - Valeant Site 28, Marietta, Georgia
  - Valeant Site 16, Buffalo Grove, Illinois
  - Valeant Site 06, Indianapolis, Indiana
  - Valeant Site 12, Overland Park, Kansas
  - Valeant Site 32, Crowley, Louisiana
  - Valeant Site 30, Clarkston, Michigan
  - Valeant Site 03, Detroit, Michigan
  - Valeant Site 20, Henderson, Nevada
  - Valeant Site 08, New York, New York
  - Valeant Site 23, Winston-Salem, North Carolina
  - Valeant Site 29, Hazleton, Pennsylvania
  - Valeant Site 24, Johnston, Rhode Island
  - Valeant Site 10, Austin, Texas
  - Valeant Site 01, Houston, Texas
  - Valeant Site 33, Port Arthur, Texas
  - Valeant Site 07, San Antonio, Texas
  - Valeant Site 13, San Antonio, Texas
  - Valeant Site 14, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tyring SK, Kircik L, Pariser DM, Woolery-Lloyd HC, Harper JC, Bhatt V, Pillai R, Guenin E. The Effects of Once-Daily Tretinoin 0.05% Lotion on Quality of Life in Patients with Moderate-to-Severe Acne Vulgaris. Am J Clin Dermatol. 2020 Dec;21(6):891-899. doi: 10.1007/s40257-020-00559-3. PMID 32886337

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized in a 1:1 ratio to receive either IDP-121(tretinoin 0.05 percent [%]) Lotion or IDP-121 Vehicle Lotion.
Groups:
- IDP-121 Lotion: IDP-121 lotion (tretinoin 0.05%) was applied topically to the face of participants with moderate to severe acne, once daily for 12 weeks.
- IDP-121 Vehicle Lotion: IDP-121 lotion vehicle was applied topically to the face of participants with moderate to severe acne, once daily for 12 weeks.
Period: Overall Study
Arm/Group | IDP-121 Lotion | IDP-121 Vehicle Lotion
Started | 413 | 407
Intent-to-treat (ITT) Population (All randomized participants who received study drug.) | 413 | 407
Safety Population (All randomized participants with ≥1 confirmed dose of study drug and ≥1 post baseline evaluation.) | 389 | 398
Completed | 342 | 364
Not Completed | 71 | 43
Not completed — Lost to Follow-up | 40 | 18
Not completed — Subject Request | 22 | 13
Not completed — Withdrawal by Parent or Guardian | 3 | 6
Not completed — Adverse Event | 3 | 0
Not completed — Noncompliance with Study Drug | 1 | 1
Not completed — Worsening Condition | 0 | 2
Not completed — Lack of Efficacy | 1 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Pregnancy | 1 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Participant ran out of study drug | 0 | 1

BASELINE CHARACTERISTICS:
Population: ITT analysis set included all randomized participants who received study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | IDP-121 Lotion | IDP-121 Vehicle Lotion | Total
Number analyzed (Participants) | 413 | 407 | 820
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.5 (7.21) | 20.7 (7.63) | 20.6 (7.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 204 | 229 | 433
  Male | 209 | 178 | 387
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 225 | 227 | 452
  Not Hispanic or Latino | 187 | 180 | 367
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 16 | 13 | 29
  Native Hawaiian or Other Pacific Islander | 1 | 3 | 4
  Black or African American | 90 | 71 | 161
  White | 297 | 311 | 608
  More than one race | 9 | 8 | 17
  Unknown or Not Reported | 0 | 0 | 0
Evaluator's Global Severity Score (EGSS) [Count of Participants; unit: Participants] — EGSS was based on a 5-point scale ranging from 0 to 4; where 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate, and 4 = severe.
  Participants
    0 - Clear | 0 | 0 | 0
    1 - Almost Clear | 0 | 0 | 0
    2 - Mild | 0 | 0 | 0
    3 - Moderate | 369 | 356 | 725
    4 - Severe | 44 | 51 | 95
Noninflammatory Lesion Count [Mean (Standard Deviation); unit: lesion count] | 46.1 (19.25) | 48.3 (19.91) | 47.2 (19.60)
Inflammatory Lesion Count [Mean (Standard Deviation); unit: lesion Count] | 26.5 (5.42) | 26.0 (5.25) | 26.2 (5.34)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in Mean Noninflammatory Lesion Count to Week 12
Description: Noninflammatory lesions were defined as follows: Open comedones (blackhead) - plugged hair follicle with dilated/open orifice, black in color; and Closed comedones (whitehead) - plugged hair follicle: small opening at skin surface. For noninflammatory facial lesions, open and closed comedones were recorded as a single count.
Time Frame: Baseline (Day 0), Week 12
Population: ITT population included all randomized participants who received study drug. Multiple imputation (Markov Chain Monte Carlo [MCMC]) was used to impute missing values.
Measure: Least Squares Mean (Standard Deviation); unit: lesion count
Arm/Group | IDP-121 Lotion | IDP-121 Vehicle Lotion
Number analyzed (Participants) | 413 | 407
lesion count | -21.9 (22.70) | -13.9 (23.30)
Statistical Analysis 1: Comparison: IDP-121 Lotion vs IDP-121 Vehicle Lotion; Analysis was performed using analysis of covariance (ANCOVA) with factors of treatment group and analysis center and the respective baseline lesion count as a covariate; Test type: Superiority; p < 0.001, ANCOVA — Threshold for significance at 0.05

2. Primary Outcome: Absolute Change From Baseline in Mean Inflammatory Lesion Count to Week 12
Description: Inflammatory lesions were defined as follows: Papule - a solid, elevated lesion less than 5 millimeters (mm); and Pustule - an elevated lesion containing pus less than 5 mm. For inflammatory facial lesions, papules and pustules were recorded as a single count, while nodular lesions were counted and recorded separately.
Time Frame: Baseline, Week 12
Population: ITT population included all randomized participants who received study drug. Multiple imputation (MCMC) was used to impute missing values.
Measure: Least Squares Mean (Standard Deviation); unit: lesion count
Arm/Group | IDP-121 Lotion | IDP-121 Vehicle Lotion
Number analyzed (Participants) | 413 | 407
lesion count | -13.9 (11.99) | -10.7 (12.12)
Statistical Analysis 1: Comparison: IDP-121 Lotion vs IDP-121 Vehicle Lotion; Analysis was performed using ANCOVA with factors of treatment group and analysis center and the respective baseline lesion count as a covariate; Test type: Superiority; p < 0.001, ANCOVA — Threshold for significance at 0.05

3. Primary Outcome: Percentage of Participants With Treatment Success at Week 12
Description: Treatment success was defined as at least a 2-grade reduction from Baseline in EGSS score and an EGSS score equating to "Clear" or "Almost Clear". EGSS was based on a 5-point scale ranging from 0 to 4; where 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate, and 4 = severe.
Time Frame: Baseline, Week 12
Population: ITT population included all randomized participants who received study drug and evaluable for EGSS score. Multiple imputation (MCMC) was used to impute missing values.
Measure: Number; unit: percentage of participants
Arm/Group | IDP-121 Lotion | IDP-121 Vehicle Lotion
Number analyzed (Participants) | 413 | 407
percentage of participants | 19.8 | 12.5
Statistical Analysis 1: Comparison: IDP-121 Lotion vs IDP-121 Vehicle Lotion; Analysis was performed using a logistic regression test (using Firth's Penalized Likelihood) with factors of treatment group and analysis center; Test type: Superiority; p = 0.007, Regression, Logistic — Threshold for significance at 0.05

4. Secondary Outcome: Percent Change From Baseline in Noninflammatory Lesion Count to Week 12
Description: as for outcome 1
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Deviation); unit: percent change
Arm/Group | IDP-121 Lotion | IDP-121 Vehicle Lotion
Number analyzed (Participants) | 413 | 407
percent change | -45.6 (44.64) | -31.9 (45.79)

5. Secondary Outcome: Percent Change From Baseline in Inflammatory Lesion Count to Week 12
Description: as for outcome 2
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Deviation); unit: percent change
Arm/Group | IDP-121 Lotion | IDP-121 Vehicle Lotion
Number analyzed (Participants) | 413 | 407
percent change | -53.4 (45.44) | -41.5 (45.68)

ADVERSE EVENTS:
Time Frame: Baseline (Day 0) up to Week 12
Description: Safety population included all randomized participants who were presumed to have used study drug at least once and who provided at least 1 post baseline evaluation.
Arm/Group | IDP-121 Lotion | IDP-121 Vehicle Lotion
All-Cause Mortality (participants affected / at risk) | 0/389 | 0/398
Serious Adverse Events (participants affected / at risk) | 2/389 | 2/398
Other Adverse Events (participants affected / at risk) | 0/389 | 0/398
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | IDP-121 Lotion (N=389) | IDP-121 Vehicle Lotion (N=398)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 2/204 | 1/229 — This is a gender-specific AE. Only female participants were at risk.
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Please contact Sponsor directly for additional information.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-07): https://cdn.clinicaltrials.gov/large-docs/56/NCT02965456/Prot_SAP_000.pdf